CLINICAL TRIAL: NCT02936648
Title: Hepatitis C Testing in VA Community-Based Outpatient Clinics (QUE 15-284)
Brief Title: Hepatitis C Testing in VA Community-Based Outpatient Clinics
Acronym: HCVCBOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QUX 16-010
Record Dates: First submitted 2016-10-11; First posted 2016-10-18 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis C
Keywords: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- quality improvement intervention (Experimental): The intervention activities included: assessment, planning, stakeholder engagement, education, ongoing process monitoring, program adaptation, problem identification and problem solving, data audit/feedback, program marketing, network development, among others.
  Interventions: Other: quality improvement intervention

INTERVENTIONS:
Other: quality improvement intervention — The intervention activities included: assessment, planning, stakeholder engagement, education, ongoing process monitoring, program adaptation, problem identification and problem solving, data audit/feedback, program marketing, network development, among others.

SUMMARY:
The VISN1 VA Hepatitis C Testing and Linkage to Care Quality Improvement project aims to increase the proportion of Veterans tested for HCV in those born between 1945-1965 and in vulnerable, high-risk groups.

DETAILED DESCRIPTION:
The VISN1 VA Hepatitis C Testing and Linkage to Care Quality Improvement project aims to: (1) increase the proportion of Veterans tested for HCV in those born between 1945-1965 and in vulnerable, high-risk groups, (2) Increase linkage to specialized HCV care among VISN 1 VA Veterans diagnosed with HCV infection, and (3) Evaluate whether race, ethnicity, gender, or other markers of social disparity influence completion of HCV testing and linkage to specialty care, and whether disparities are reduced by the planned VISN 1 VA HCV Quality Improvement (QI) program. The central focus is to reduce delays in diagnosis and linkage to treatment evaluation, management of comorbidities and contraindications, and subsequent initiation.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* Born in the period of 1945-1965 ("birth cohort")
* With an outpatient visit in primary care at a VISN1 facility in FY 2016

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2209 (Actual)
Dates: Start 2015-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen L. Gifford, MD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA; Mari-Lynn Drainoni, PhD, Principal Investigator — Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA
Locations (1):
- Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yakovchenko V, DeSotto K, Drainoni ML, Lukesh W, Miller DR, Park A, Shao Q, Thornton DJ, Gifford AL. Using Lean-Facilitation to Improve Quality of Hepatitis C Testing in Primary Care. J Gen Intern Med. 2021 Feb;36(2):349-357. doi: 10.1007/s11606-020-06210-5. Epub 2020 Sep 15. PMID 32930938

RESULTS

PARTICIPANT FLOW:
Groups:
- Quality Improvement Intervention: quality improvement Intervention
  quality improvement : HCV Testing quality improvement
Period: Overall Study
Arm/Group | Quality Improvement Intervention
Started | 2209
Completed | 2209
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Number of veterans with an outpatient primary care visit in the month.
Groups:
- Baseline Characteristics at Intervention Sites: QI Intervention. QI: HCV Testing QI. Baseline characteristics at intervention sites, pre-implementation.
Arm/Group | Baseline Characteristics at Intervention Sites
Number analyzed (Participants) | 2209
Age, Customized [Count of Participants; unit: Participants]
  Age: <60 | 505
  Age: >60 | 1704
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136
  Male | 2073
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 1526
  Unknown or Not Reported | 654
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 56
  White | 1470
  More than one race | 0
  Unknown or Not Reported | 683

OUTCOME MEASURES:

1. Primary Outcome: HCV Antibody Test
Description: Number of Participants with HCV Antibody Test
Time Frame: within 30 days of outpatient primary care visit
Measure: Count of Participants; unit: Participants
Groups:
- Quality Improvement Intervention: QI Intervention
  QI: HCV Testing QI
Arm/Group | Quality Improvement Intervention
Number analyzed (Participants) | 2209
Participants | 574

ADVERSE EVENTS:
Groups:
- HCV Testing QI: Intervention/HCV Testing QI: lean and facilitation implementation to increase HCV testing
Arm/Group | HCV Testing QI
All-Cause Mortality (participants affected / at risk) | 0/2209
Serious Adverse Events (participants affected / at risk) | 0/2209
Other Adverse Events (participants affected / at risk) | 0/2209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes